CLINICAL TRIAL: NCT05976620
Title: Clinical Study of 18F Labeled Probe Targeting Fibroblast Activation Protein Inhibitor and Integrin avβ3 (FAPI-RGD) in Breast Tumors
Brief Title: Clinical Study of 18F-FAPI-RGD in Breast Tumors
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-Breast cancer
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Breast Tumors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the value of 18F-FAPI-RGD PET/CT imaging in Breast Tumors. Participants will undergo clinical evaluation and 18F-FAPI-RGD PET/CT examination.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant disease in women worldwide.Early detection, accurate diagnosis and staging are the keys to effective treatment for breast cancer patients.18F-FDG PET/CT has become an important imaging method for the diagnosis and staging of breast cancer.However,FDG PET has certain limitations, including false-positive uptake for acute and chronic infections and false-negative uptake for less aggressive histological subtypes of breast cancer.In a number of studies, 68Ga-FAPI PET was positively correlated with the pathological grade and end-stage of primary breast cancer lesions, and SUVmax could predict tumor grade, final stage and lymph node metastasis. Compared with 18F-FDG,68Ga-FAPI PET/CT had higher specificity and accuracy in judging lymph node metastasis.Integrin αvβ3 is highly expressed in neovascular endothelial cells and tumor cells including breast cancer, and plays an important role in regulating tumor growth, angiogenesis, local invasion and metastasis potential.The use of integrin αvβ3 specific imaging probes derived from RGD peptides in breast cancer patients has also been reported.

Several studies have confirmed that the heterodimer is superior to the corresponding monomer due to the polyvalent effect, thus improving the binding affinity and increasing the number of effective receptors.In order to simultaneously target FAP and integrin αvβ3, we synthesized the heterodimeric peptide FAPI-RGD from FAPI and RGD.FAPI-RGD is a heterodimeric peptide that targets FAP and αvβ3-integrin receptors. 68Ga-FAPI-RGDPET/CT imaging has been used in clinical imaging studies in patients with a variety of tumors.Therefore, we plan to use 18F-FAPI-RGD PET/CT imaging for the diagnosis and treatment of breast cancer, and preliminary experiments have confirmed that this examination has a good imaging effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* No gender difference
* Patients who have been diagnosed with, or are clinically highly suspected of, breast tumors and have had no other treatment within 3 months
* Tumor size (T), lymph node status (N), and overall clinical stage of diagnosed patients were determined according to the American Joint Committee on Cancer criteria revised in 2010

Exclusion Criteria:

* Patients with a second primary tumor
* Pregnant or breastfeeding
* Severe liver or kidney disease
* Claustrophobia or other PET/CT scan contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed or highly suspected breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Correlation between clinical indicators and PET/CT results | 2 months
  Correlation of Immunohistochemical indexes, ultrasound, X-ray, CT, MRI, tumor markers，estrogen assay and 18F-FAPI-RGD PET/CT results

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China